CLINICAL TRIAL: NCT02259049
Title: The Effects of L-Tyrosine on Non-invasive Ambulatory Blood Pressure and Heart Rate Monitoring in Parkinson's Disease
Brief Title: The Effects of L-Tyrosine on 24 Hour Blood Pressure and Heart Rate in Parkinson's Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Associate Professor, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BHS-1056
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2014-09

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Tyrosine; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Tyrosine (Active Comparator): We will administer 1,000 mg of L-tyrosine BID for 24 hours and record BP and HR.
  Interventions: Dietary Supplement: L-tyrosine; Dietary Supplement: Sugar Pill
- Sugar Pill (Placebo Comparator): We will administer a sugar pill BID for 24 hours and record BP and HR.
  Interventions: Dietary Supplement: L-tyrosine; Dietary Supplement: Sugar Pill

INTERVENTIONS:
Dietary Supplement: L-tyrosine — Each subject will receive 2,000 mg of L-tyrosine BID for 24 hours.
Dietary Supplement: Sugar Pill — Each subject will receive a sugar pill BID for 24 hours.

SUMMARY:
The investigators are observing the effects 2,000 mg of L-tyrosine will have on 24 hour blood pressure fluctuations in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
We will be monitoring 24 hour ambulatory BP and HR in subjects with PD on 3 separate visits. The first visit will be without an intervention to establish a baseline of 24 hour BP fluctuations. One week later the subject will be given either L-tyrosine (2,000 mg) with B6 (10 mg) or a sugar pill. We will monitor 24 hour BP and HR after supplementation. One week later the subject will repeat the same procedures with either supplement or placebo.

This is a total of 3 visits with 24 hour ambulatory BP and HR monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have a diagnosis of PD by a licensed neurologist according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (UKPDBB).(Goetz, 2010) The UKPDBB is a 3 step diagnostic tool which defines inclusion and exclusion criteria for diagnosing PD
2. between 35 and 79 years of age
3. mentally able to participate in the study

Exclusion Criteria:

1. Pregnancy
2. any person who is currently taking amino acid supplements.
3. Any history of myocardial infarction, stent, or CABG
4. Phenylketonurics
5. Untreated hypertension

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 24 hours

SECONDARY OUTCOMES:
Heart Rate | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, PhD, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States